CLINICAL TRIAL: NCT03749447
Title: An Extended Access Program to Assess Long Term Safety of Bardoxolone Methyl in Patients With Chronic Kidney Disease
Brief Title: An Extended Access Program for Bardoxolone Methyl in Patients With CKD (EAGLE)
Acronym: EAGLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinuation of all bardoxolone chronic kidney disease programs
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-1803; 2018-003253-24 (EudraCT Number)
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Diseases; Alport Syndrome; Autosomal Dominant Polycystic Kidney
Keywords: Bardoxolone methyl; CDDO-ME; RTA 402; Alport Syndrome; Autosomal Dominant Polycystic Kidney; ADPKD
MeSH Terms: conditions — Renal Insufficiency, Chronic; Nephritis, Hereditary; Polycystic Kidney, Autosomal Dominant | interventions — bardoxolone methyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bardoxolone methyl (Experimental): Adult participants received bardoxolone methyl capsules, once daily (QD) at a starting dose of 5 milligrams (mg), followed by dose- escalation to 10 mg at Week 2 (Day 14 ± 3), and to 20 mg at Week 4 (Day 28 ± 3). Based on the eligibility UACR >300 milligrams per gram (mg/g), the dose was increased to 30 mg starting from Week 6 (Day 42 ± 3) until the end of the study.
  Participants under 18 years of age received bardoxolone methyl capsules at a starting dose of 5 mg every other day during the first week and QD during the second week of the study, followed by dose-escalation to 10 mg at Week 2 and to 20 mg at Week 4. Based on the eligibility UACR >300 mg/g, the dose was increased to 30 mg starting from Week 6 until the end of the study.
  Interventions: Drug: Bardoxolone methyl

INTERVENTIONS:
Drug: Bardoxolone methyl — Bardoxolone methyl capsules
  Other Names: RTA 402

SUMMARY:
This extended access study will assess the long-term safety and tolerability of bardoxolone methyl in qualified patients with chronic kidney disease (CKD) who previously participated in one of the qualifying clinical studies with bardoxolone methyl. Patients will remain in the study until bardoxolone methyl is available through commercial channels or until patient withdrawal, whichever is sooner.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are participating (or who have participated) in qualifying studies and who have not been required to discontinue study treatment for protocol or safety reasons and who have completed required End-of-Treatment and/or Follow-up visits in a prior clinical study with bardoxolone methyl and who, according to the assessment of the investigator, have a potential positive benefit-risk assessment for participating in the trial.
* Meets the following eligibility criteria based on assessments from the prior qualifying study (last on-treatment visit) or from a screening visit, if applicable:

  1. Not expected to reach end stage kidney disease (ESKD) or nephrotic syndrome within 12 weeks of study enrollment, in the investigator's judgement; subjects with eGFR <20 ml/min/1.73m2 should be discussed with the medical monitor before enrollment (e.g., such subjects with an average rate of eGFR decline > 1.0 ml/min/1.73m2 per month in the 3 months prior to eligibility assessment may not be eligible);
  2. BNP < 200 pg/mL at the last on-treatment visit in the prior qualifying study or at a new screening visit, if applicable;
  3. No occurrence of a cardiovascular serious adverse event in the prior qualifying study or in the interval between the end of the qualifying study and the screening visit, if applicable.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Evidence of a personally signed and dated informed consent document (and assent form if necessary) indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study prior to initiation of any protocol-mandated procedures.

Exclusion Criteria:

* Participation in other investigational clinical studies involving interventional products being tested or used in a way different from the approved form or when used for an unapproved indication;
* Patients who have an ongoing SAE from a clinical study that is assessed by the investigator as related to bardoxolone methyl;
* Unwilling to practice acceptable methods of birth control (both males who have partners of childbearing potential and females of childbearing potential) while screening, taking study drug and 30 days after the last study drug dose;
* Women who are pregnant or breastfeeding;
* Patient is, in the opinion of the investigator, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason;
* Known hypersensitivity to any component of the study drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (87):
- United States (61):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Apogee Clinical Research, Huntsville, Alabama
  - Arizona Kidney Disease and Hypertension Research Services, PLLC, Glendale, Arizona
  - Centricity Research Phoenix Multispecialty, Mesa, Arizona
  - California Institute Renal Research, La Mesa, California
  - Academic Medical Research Institute, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Apex Research of Riverside, Riverside, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco - Children's Renal Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Western Nephrology, Arvada, Colorado
  - University of Colorado Anschutz Medical Center, Aurora, Colorado
  - Colorado Kidney Care, PC, Denver, Colorado
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Innovation Medical Research, Inc., Palmetto Bay, Florida
  - USF Health South Tampa Center, Tampa, Florida
  - Florida Premier Research Institute, LLC, Winter Park, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Boise Kidney & Hypertension, PLLC, Caldwell, Idaho
  - Boise Kidney & Hypertension, PLLC, Meridian, Idaho
  - Northwestern University, Chicago, Illinois
  - Nephrology Research NorthShore University Health System, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - The Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center - Division of Nephrology, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Nephrology Center, PC, Kalamazoo, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - KSOSN, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Mountain Kidney & Hypertension Associates, Asheville, North Carolina
  - North Carolina Nephrology, Cary, North Carolina
  - Metrolina Nephrology Associates, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Metrolina Nephrology Associates, Gastonia, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Remington-Davis Clinical Research, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - South Carolina Nephrology & Hypertension Center, Inc, Orangeburg, South Carolina
  - Arlington Nephrology, Arlington, Texas
  - Research Management, Inc., Austin, Texas
  - Renal Disease Research Institute, Dallas, Texas
  - DaVita Med Center, Houston, Texas
  - Southwest Houston Research, Houston, Texas
  - Clinical Advancement Center, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Nephrology Associates of Northern Virginia, Inc., Fairfax, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Milwaukee Nephrologists, SC, Wauwatosa, Wisconsin
- Australia (4):
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Melbourne Renal Research Group, Reservoir, Victoria
  - The Royal Melbourne Hospital, Parkville
- France (2):
  - Chu Grenoble Alpes, Grenoble
  - Hopital Necker, Universite Paris Descartes, Paris
- Japan (17):
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Toranomon Hospital Kajigaya, Kawasaki, Kanagawa
  - St Marianna University Hospital, Kawasaki, Kanagawa
  - JCHO Sendai Hospital, Sendai, Miyagi
  - Kitano Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - Saitama Children's Medical Center, Saitama-shi, Saitama
  - Juntendo University Hospital, Bunkyō-Ku, Tokyo
  - Jutendo University Hospital, Bunkyō-Ku, Tokyo
  - Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - Toranomon Hospital, Minato-Ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku, Tokyo
  - Niigata University Medical and Dental Hospital, Niigata
  - Local Incorporated Administrative Agency Osaka City Hospital Organization Osaka City General Hospital, Osaka
- Puerto Rico Clinical and Translational Research Consortium (PRCTRC), Rio Piedras, Puerto Rico
- Spain (2):
  - Fundacio Puigvert, Barcelona, Catalonia
  - Hospital Virgen de la Arrixaca, El Palmar, Murcia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the investigative sites in the United States, Australia, Japan, Spain, Puerto Rico and France from 08 March 2019 to 23 August 2023.
Pre-assignment Details: A total of 270 eligible participants who participated in the previous qualifying studies i.e., 402-C-1603 (NCT03019185) and 402-C-1808 (NCT03918447) of bardoxolone methyl were enrolled in this study. Data was summarized as per the treatment received in the previous qualifying studies.
Groups:
- Prior Placebo to Bardoxolone Methyl: Participants who received placebo in the previous qualifying studies, 402-C-1603 (NCT03019185) or 402-C-1808 (NCT03918447), and received bardoxolone methyl in this study.
  Adult participants received bardoxolone methyl capsules, once daily (QD) at a starting dose of 5 milligrams (mg), followed by dose- escalation to 10 mg at Week 2 (Day 14 ± 3), and to 20 mg at Week 4 (Day 28 ± 3). Based on the eligibility urine albumin to creatinine ratio (UACR) >300 milligrams per gram (mg/g), the dose was increased to 30 mg starting from Week 6 (Day 42 ± 3) until the end of the study.
  Participants under 18 years of age received bardoxolone methyl capsules at a starting dose of 5 mg every other day during the first week and QD during the second week of the study, followed by dose-escalation to 10 mg at Week 2 and to 20 mg at Week 4. Based on the eligibility UACR >300 mg/g, the dose was increased to 30 mg starting from Week 6 until the end of the study.
- Prior Bardoxolone Methyl to Bardoxolone Methyl: Participants who received bardoxolone methyl in the previous qualifying studies, 402-C-1603 (NCT03019185) or 402-C-1808 (NCT03918447), and received bardoxolone methyl in this study.
  Adult participants received bardoxolone methyl capsules, QD at a starting dose of 5 mg, followed by dose-escalated to 10 mg at Week 2 (Day 14 ± 3), and to 20 mg at Week 4 (Day 28 ± 3). Based on the eligibility UACR >300 mg/g, the dose was increased to 30 mg starting from Week 6 (Day 42 ± 3) until the end of the study.
  Participants under 18 years of age received bardoxolone methyl capsules at a starting dose of 5 mg every other day during the first week and QD during the second week of the study, followed by dose-escalation to 10 mg at Week 2 and to 20 mg at Week 4. Based on the eligibility UACR >300 mg/g, the dose was increased to 30 mg starting from Week 6 until the end of the study.
Period: Overall Study
Arm/Group | Prior Placebo to Bardoxolone Methyl | Prior Bardoxolone Methyl to Bardoxolone Methyl
Started | 143 | 127
Completed | 0 | 0
Not Completed | 143 | 127
Not completed — Adverse Event | 11 | 3
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Reason Not Specified | 0 | 3
Not completed — Physician Decision | 4 | 3
Not completed — Protocol-Specified Withdrawal Criteria Met | 1 | 3
Not completed — Study Terminated By Sponsor | 112 | 105
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Non-compliance With Study Drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who had received at least 1 dose of bardoxolone methyl in the 402-C-1803 study.
Groups:
- Prior Placebo to Bardoxolone Methyl: Participants who received placebo in the previous qualifying studies, 402-C-1603 (NCT03019185) or 402-C-1808 (NCT03918447), and received bardoxolone methyl in this study.
  Adult participants received bardoxolone methyl capsules, QD at a starting dose of 5 mg, followed by dose- escalation to 10 mg at Week 2 (Day 14 ± 3), and to 20 mg at Week 4 (Day 28 ± 3). Based on the eligibility UACR >300 mg/g, the dose was increased to 30 mg starting from Week 6 (Day 42 ± 3) until the end of the study.
  Participants under 18 years of age received bardoxolone methyl capsules at a starting dose of 5 mg every other day during the first week and QD during the second week of the study, followed by dose-escalation to 10 mg at Week 2 and to 20 mg at Week 4. Based on the eligibility UACR >300 mg/g, the dose was increased to 30 mg starting from Week 6 until the end of the study.
- Total: Total of all reporting groups
Arm/Group | Prior Placebo to Bardoxolone Methyl | Prior Bardoxolone Methyl to Bardoxolone Methyl | Total
Number analyzed (Participants) | 143 | 127 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (13.26) | 48.3 (13.82) | 48.6 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 78 | 166
  Male | 55 | 49 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 2 | 0 | 2
  Race: Asian | 17 | 16 | 33
  Race: Black or African American | 9 | 9 | 18
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: White | 112 | 96 | 208
  Race: Other | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic/Latino | 15 | 12 | 27
  Ethnicity: Non-Hispanic/Latino | 128 | 115 | 243

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is a medically important event. AEs and SAEs that occurred within 30 days after the last dose were considered treatment-emergent. The study follow-up assessment was collected within 14 to 35 days after the last dose.
Time Frame: From the first dose of the study drug (baseline) up to the end of the study follow-up (up to 4.2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Placebo to Bardoxolone Methyl | Prior Bardoxolone Methyl to Bardoxolone Methyl
Number analyzed (Participants) | 143 | 127
Participants
  AEs | 128 | 105
  SAEs | 12 | 20

ADVERSE EVENTS:
Time Frame: From the first dose of the study drug (baseline) up to the end of the study follow-up (up to 4.2 years)
Description: The safety population included all participants who had received at least 1 dose of bardoxolone methyl in the 402-C-1803 study.
Arm/Group | Prior Placebo to Bardoxolone Methyl | Prior Bardoxolone Methyl to Bardoxolone Methyl
All-Cause Mortality (participants affected / at risk) | 1/143 | 1/127
Serious Adverse Events (participants affected / at risk) | 12/143 | 20/127
Other Adverse Events (participants affected / at risk) | 127/143 | 104/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Placebo to Bardoxolone Methyl (N=143) | Prior Bardoxolone Methyl to Bardoxolone Methyl (N=127)
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Biopsy kidney (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Placebo to Bardoxolone Methyl (N=143) | Prior Bardoxolone Methyl to Bardoxolone Methyl (N=127)
Anaemia (Blood and lymphatic system disorders) | 9 | 6
Nausea (Gastrointestinal disorders) | 12 | 13
Diarrhoea (Gastrointestinal disorders) | 16 | 8
Abdominal pain (Gastrointestinal disorders) | 9 | 5
Fatigue (General disorders) | 14 | 8
Oedema peripheral (General disorders) | 10 | 11
Pyrexia (General disorders) | 7 | 7
Corona virus infection (Infections and infestations) | 22 | 27
Upper respiratory tract infection (Infections and infestations) | 12 | 12
Nasopharyngitis (Infections and infestations) | 5 | 8
Sinusitis (Infections and infestations) | 5 | 8
Alanine aminotransferase increased (Investigations) | 37 | 8
Aspartate aminotransferase increased (Investigations) | 24 | 7
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 13 | 11
Brain natriuretic peptide increased (Investigations) | 11 | 5
Gamma-glutamyltransferase increased (Investigations) | 11 | 0
Blood creatinine increased (Investigations) | 3 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 57 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 7
Headache (Nervous system disorders) | 16 | 9
Dizziness (Nervous system disorders) | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Hypertension (Vascular disorders) | 8 | 9
Urinary tract infection (Infections and infestations) | 8 | 12

LIMITATIONS AND CAVEATS:
Early termination of trial due to discontinuation of all bardoxolone chronic kidney disease programs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT03749447/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT03749447/SAP_001.pdf